CLINICAL TRIAL: NCT03495960
Title: Randomized Phase II Trial on Fitness- and Comorbidity- Tailored Treatment in Elderly Patients With Newly Diagnosed Primary CNS Lymphoma (FIORELLA Trial)
Brief Title: Study on Tailored Treatment in Elderly Patients With Newly Diagnosed Primary Lymphoma of Central Nervous System
Acronym: FIORELLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG45
Record Dates: First submitted 2018-03-23; First posted 2018-04-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: non-Hodgkin's lymphoma; elderly; PCNSL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Methotrexate; Procarbazine; Lenalidomide; Radiotherapy; Temozolomide

STUDY DESIGN:
Intervention Model Description: Multicenter open label phase II trial. The patients will be stratified according to their suitability to tolerate an induction chemo-immunotherapy regimen containing high-dose methotrexate.
  Patients eligible for high-dose methotrexate-based induction chemotherapy will enter the run-in phase of Part A of the study and after the induction phase will be randomly assigned to procarbazine or lenalidomide maintenance monotherapy. Forty assessable patients per treatment arm are required.
  Patients ineligible for high-dose methotrexate-based induction chemotherapy will be treated în Part B with concomitant whole-brain radiotherapy, temozolomide and rituximab and will receive temozolomide as maintenance.According to the Simon's two-stage minimax design, 46 patients will be treated in the first stage. If ≤ 16 patients will be progression-free at 2 years from maintenance treatment start, the study will be stopped. Otherwise, 19 additional patients will be treated for a total of 65
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lenalidomide (experimental arm of part A) (Experimental): Patients in part A will receive 2 courses of induction chemo-immunotherapy:
  Rituximab 375 mg/m2 i.v. on days -6, 1, 15, 29; Methotrexate 3 g/m2 0.5 g/m2 in 15 min. +2.5 g/m2 in 3-hr inf. on days 2,16,30; Procarbazine 60 mg/m2/d oral on days 2 to 11.
  The duration of each treatment course is 43 days. Patients will then be randomized to receive lenalidomide or procarbazine as maintenance therapy.
  Lenalidomide is given 25 mg/d per os, days 1 to 21 every 4 weeks for 24 courses
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Procarbazine; Drug: Lenalidomide
- Procarbazine (comparator arm of part A) (Active Comparator): Patients in part A will receive 2 courses of induction chemo-immunotherapy:
  Rituximab 375 mg/m2 i.v. on days -6, 1, 15, 29; Methotrexate 3 g/m2 0.5 g/m2 in 15 min. +2.5 g/m2 in 3-hr inf. on days 2,16,30; Procarbazine 60 mg/m2/d oral on days 2 to 11.
  The duration of each treatment course is 43 days. Patients will then be randomized to receive lenalidomide or procarbazine as maintenance therapy.
  Procarbazine is given 100 mg/d per os, days 1 to 5 every 4 weeks for 6 courses
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Procarbazine
- Radiotherapy, temozolomide and rituximab (single arm part B) (Other): Patients ineligible for high-dose-methotrexate will be treated in the single-arm phase II part B of the trial and will receive
  * whole-brain radiotherapy (2340 cGy in 5 weekly fractions)
  * temozolomide 75 mg/m2/d during radiotherapy
  * 4 weekly doses of rituximab 375 mg/m2, starting on day 2 of the whole-brain radiotherapy.
  Patients will then receive maintenance therapy with 12 courses of temozolomide administered on days 1-5, every 4 weeks at a dose of 150 mg/m2/d at the first course, and of 200 mg/m2/d at the subsequent courses.
  Interventions: Drug: Rituximab; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Rituximab — PART A - INDUCTION PHASE During the primary chemo-immunotherapy (PRIMAIN regimen, 2 courses; every 43 days) administered as induction in the PART A of the study, Rituximab is given 375 mg/m2 as standard infusion at days -6, 1, 15 & 29. Rituximab on day -6 will be delivered only during the first course; it will be delivered between day -6 and day 0 according to clinical requirements and patient's conditions. Some patients would need for a fast chemotherapy starting.
  PART B - INDUCTION PHASE Patients ineligible for high-dose methotrexate, will be assigned to receive concomitant whole brain radiotherapy-temozolomide-rituximab (Induction Part B). Rituximab is given 375 mg/m2 in 4 weekly doses, starting on day 2 of radiotherapy.
Drug: Methotrexate — During the primary chemo-immunotherapy (PRIMAIN regimen, 2 courses; every 43 days) administered as induction in the PART A of the study, Methotrexate is given 3 g/m2 as infusion (0.5 g/m2 in 15 min. + 2.5 g/m2 in 3-hr infusion) on days 2, 16 & 30
  Arms: Lenalidomide (experimental arm of part A); Procarbazine (comparator arm of part A)
Drug: Procarbazine — PART A - INDUCTION PHASE During the primary chemo-immunotherapy (PRIMAIN regimen, 2 courses; every 43 days) administered as induction in the PART A of the study, Procarbazine is given oral 60 mg/m2/d from days 2 to 11
  PART A - MANTEINANCE PHASE (control arm) Patients responsive or with stable disease after two courses of PRIMAIN regimen (the induction treatment) will be randomly allocated to receive two different maintenance therapies. Maintenance will start on day 60 of the 2nd PRIMAIN course.
  Procarbazine represents the control arm and is given oral 100 mg/d from day 1 to 5 for 6 courses, every 4 weeks.
  Arms: Lenalidomide (experimental arm of part A); Procarbazine (comparator arm of part A)
Drug: Lenalidomide — Patients responsive or with stable disease after two courses of PRIMAIN regimen (the induction treatment) will be randomly allocated to receive two different maintenance therapies. Maintenance will start on day 60 of the 2nd PRIMAIN course.
  Lenalidomide represents the experimental arm and is given oral 25 mg/d from day 1 to 21 for 24 courses; every 4 weeks.
  Arms: Lenalidomide (experimental arm of part A)
Radiation: Radiotherapy — Patients ineligible for high-dose methotrexate, will be assigned to receive concomitant whole brain radiotherapy-temozolomide-rituximab (Induction Part B). Whole-brain will be irradiated by two opposite lateral fields including the first two cervical vertebras and the posterior two thirds of the eyes. Photons of 4 - 10 MeV, 180 - 200 cGy per day, 5 weekly fractions will be employed
  Arms: Radiotherapy, temozolomide and rituximab (single arm part B)
Drug: Temozolomide — PART B - INDUCTION PHASE Patients ineligible for high-dose methotrexate, will be assigned to receive concomitant whole brain radiotherapy-temozolomide-rituximab (Induction Part B). Temoyolomide is given 75 mg/m2/d, every day for the whole duration of radiotherapy.
  PART B - MAINTENANCE PHASE Temozolomide is also given as maintenance in Part B. The treatment consists of 12 courses where temozolomide is administered on days 1-5, every 4 weeks at a dose of 150 mg/m2/d at the first course, and of 200 mg/m2/d at the subsequent courses,
  Arms: Radiotherapy, temozolomide and rituximab (single arm part B)

SUMMARY:
Primary central nervous system lymphomas are rare aggressive malignancies, usually treated in two steps: an induction phase (where a combination of chemotherapy is given) followed by a consolidation phase (where patients usually receive one of the following: whole-brain irradiation, chemotherapy supported by autologous stem-cell transplantation, other type of chemotherapy, or are just observed).

The feasibility of this overall strategy, for several reasons, is limited in elderly patients .

This study involves patients aged ≥70 years. The more fit patients will receive the standard chemotherapy combination (high-dose methotrexate, procarbazine and rituximab) as induction. Responding patients will receive either procarbazine or lenalidomide as maintenance therapy; the aim is to evaluate the efficacy of these two drugs.

The more fragile patients will receive a less aggressive therapy consisting of concomitant whole-brain radiotherapy, temozolomide and rituximab as induction therapy, followed by temozolomide as maintenance treatment; the aim is to evaluate the efficacy of this combination of treatment.

DETAILED DESCRIPTION:
Primary central nervous system lymphomas (PCNSL) are rare aggressive malignancies, mostly of B-cell origin, representing 4% of intracranial neoplasms and 4-6% of extranodal non-Hodgkin's lymphomas (NHL). Despite improvements in treatment, PCNSL is associated with an aggressive course and unsatisfactory outcome. The median age at diagnosis is 61 years and age over 60 years has been reported to be an independent factor for a poorer outcome.

The modern treatment of PCNSL includes two phases: induction and consolidation. The induction phase usually consists of a polychemotherapy combination, including high-dose methotrexate as a critical drug, while there are at least four different strategies that can be used as consolidation: whole-brain irradiation, myeloblative chemotherapy supported by autologous stem-cell transplantation, non-myeloblative chemotherapy, observation (only in patients who achieve complete remission after induction).

The feasibility of this overall strategy is limited, for several reasons, in elderly patients with newly diagnosed PCNSL. High-doses of antimetabolite-based chemotherapy, the standard induction for patients younger than 70 years, is often not feasible in elderly patients. Among maintenance strategies, simple observation results in unacceptably high relapse rate and associated mortality while whole-brain irradiation and aggressive chemotherapies are associated with unacceptable toxicity and poor outcome. Thus, new strategies aimed at obtaining durable responses with an acceptable tolerability and reduced risk of neurocognitive decline are needed and these strategies should be tailored not only based on the patients' age but also on their specific co-morbidities and general health conditions.

For the present trial, all patients aged ≥70 years taken into care at the participating sites will be invited to participate and after informed consent signature their baseline data will be collected in the trial database, including data of patients resulting in screening failure. This will allow to verify any potential screening bias by comparing the characteristics of included and excluded patients. Patients fulfilling the eligibility criteria are then screened for their suitability to receive a more or less aggressive anticancer treatment and assigned to two different treatment strategies accordingly.

Part A:

The more fit patients are assigned to the trial Part A and will receive the standard combination of high-dose methotrexate, procarbazine and rituximab as induction. Responding patients will subsequently be randomized to receive either procarbazine or lenalidomide as maintenance therapy.

Procarbazine is a lipophilic oral alkylating agent, easily crossing the blood brain barrier (up to 100% of plasma levels). There is no known cumulative toxicity for procarbazine and it is therefore currently in use as a viable maintenance treatment option aimed at eliminating residual lymphoma cells in the CNS and reduce the risk of relapse. Lenalidomide is an oral immunomodulatory agent, active against diffuse large B cell lymphoma, the most common category in PCNSL, which can be taken for years, showing an excellent safety profile. On this background, the Part A of the present trial consists of a randomized phase II trial conducted in elderly patients with newly diagnosed PCNSL responsive to high-dose methotrexate-based chemotherapy, comparing two different maintenance strategies: the oral chemotherapeutic drug procarbazine and the oral immunomodulatory agent lenalidomide.

Part B:

The more fragile patients are assigned to the trial Part B and will receive a less aggressive therapy consisting of concomitant whole-brain radiotherapy, temozolomide and rituximab as induction therapy, followed by temozolomide single-agent as maintenance treatment.

Whole-brain radiotherapy is the main therapeutic choice for patients with contraindications to chemotherapy and in particular for elderly patients. Brain irradiation is usually associated with transient disruption of the blood-tumor barrier, occurring from 1 week after the initiation of radiotherapy to 1 month after its completion, during which pharmaceutical agents have maximum access to tumor tissue. Concomitant delivery of active cytostatics, therefore, could result in increased tumor uptake. Concomitant delivery of radiotherapy and temozolomide is currently used as standard approach for the treatment of high-grade gliomas, with acceptable toxicity despite the use of a larger irradiation dose. Based on the above, in the Part B of the present trial, temozolomide and rituximab, two agents active against PCNSL, are delivered concomitantly to whole-brain radiotherapy to obtain a synergistic effect of radiation damage, antineoplastic effect of rituximab and cytostatic and radiomimetic effects of temozolomide. Finally, temozolomide maintenance has shown to be beneficial regarding sustained remission after initial response to induction therapy and its suitability to improve disease control in responding patients not fit for more aggressive therapies will therefore be tested in the Part B of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically assessed diagnosis of CD20+ diffuse large B-cell lymphoma.
* Diagnostic sample obtained by stereotactic or surgical biopsy, CSF cytology examination or vitrectomy.
* Lymphoma exclusively localized in the central nervous system (brain parenchyma and/or meningeal/CSF dissemination and/or eyes and/or cranial nerves).
* Previously untreated patients (previous or ongoing steroid therapy admitted).
* Age ≥70 years
* Patients not eligible for high-dose chemotherapy supported by autologous stem cell transplant
* ECOG PS ≤3.
* Adequate bone marrow, cardiac, renal, and hepatic function
* No previous or concurrent malignancies with the exception of surgically cured carcinoma in-situ of the cervix, carcinoma of the skin or other cancers without evidence of disease at least for 3 years (patients with a previous lymphoma at any time are NOT eligible).
* Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* No concurrent treatment with other experimental drugs.
* Patients receiving oral lenalidomide or procarbazine must agree to avoid sharing the study medication with another person and to return all unused study drug to the investigator.
* Male patients must agree to always use a latex or synthetic condom during any sexual contact with females of reproductive potential while taking lenalidomide, during dose interruptions and for up to 7 days after treatment discontinuation, even if they have undergone a successful vasectomy.
* Informed consent from the patient, or legal representative, obtained before registration.

Exclusion Criteria:

* Lymphoma entity other than diffuse large B-cell lymphoma.
* Extra-CNS disease.
* Lymphoma exclusively localized in the eyes
* Lymphoma infiltration of the cranial nerves as exclusive site of disease
* Previous antineoplastic treatment for the PCNSL.
* Patients eligible for ASCT.
* HBsAg- and HCV-positive patients; HBsAg- and HCV-positive patients. HBcAb+ is not exclusion criteria in the absence of detectable levels HBVDNA.
* HIV disease or immunodeficiency.
* Severe concomitant illnesses/medical conditions (e.g. impaired respiratory and/or cardiac function, uncontrolled diabetes mellitus despite optimal medical management).
* Active infectious disease.
* Hypersensitivity to any active principle and/or any excipient according to the contraindications reported in the Summary of Product Characteristics (SmPCs) of the anticancer drugs used in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Two years Progression Free Survival (PFS) - part A | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  The primary objective is to evaluate whether lenalidomide administered as maintenance treatment after achievement of disease stabilization or better response by standard induction therapy results in a higher 2-year PFS rate as compared to procarbazine maintenance.
  The corresponding primary endpoint is the difference in 2-years PFS between the two treatment arms.
Two years Progression Free Survival (PFS) - part B | From date of maintenance start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
Duration of response (part A) | From date of first assessment of response (PR or CR) until the date of first documented progression, assessed up to 2 years from randomization.
  Difference between the two arms in time from first assessment of response (PR or CR) to relapse/progression
Response Rates (part B) | From the start of the treatment until disease progression, assessed up to 2 years from start of maintenance.
  Proportion of patients showing CR, PR, SD, PD as best response to treatment
Overall survival (OS) | From date of induction treatment start until the date of death from any cause or the date of the last visit in patients still alive at study end, assessed up to 2 years from start of maintenance.
Relapse rates and patterns | From the start of the treatment until disease progression, assessed up to 2 years from start of maintenance.
  Analysis of the following relapse rates and patterns: primary site vs. secondary CNS sites vs. extra-CNS sites; CNS sites: brain, meninges, cranial nerves, and/or eyes
Incidence of Treatment-Emergent Adverse Events | From the 2 weeks preceding treatment start through study completion, an average of 2.5 years
  Analysis of adverse events and adverse reactions incidence and severity
Early and late neurotoxicity | From maintenance up to 2 years.
  Analysis of incidence and severity of early and late neurotoxicity assessed by specific neuropsychological and quality of life tests up to 2 years from maintenance treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Andrès JM Ferreri, MD, Study Chair — IRCCS San Raffaele Scientific Institute, Milan, Italy
Locations (34):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- Finland (2):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Italy (25):
  - Centro di Riferimento Oncologico, Aviano, (PN)
  - Ospedale C.e G. Mazzoni, Ascoli Piceno
  - Bari IRCCS Istituto Tumori, Bari
  - ASST Spedali Civili di Brescia, Brescia
  - Ospedale Antonio Perrino, Brindisi
  - Azienda Ospedaliera Universitaria (AOU) Careggi, Florence
  - Meldola, IRST - ISTITUTO SCIENTIFICO ROMAGNOLO PER LO STUDIO E LA CURA DEI TUMORI, Meldola
  - Milano, IRCCS Ospedale San Raffaele, Milan
  - Milano - Îstituto Besta, Milan
  - Milano Niguarda, Milan
  - Modena, Policlinico Universitario, Modena
  - ASST Monza - Ospedale S. Gerardo, Monza
  - Pescara, Presidio Ospedaliero UOS dipartimentale centro di diagnosi e terapia Linfomi, Pescara
  - Piacenza, Piacenza
  - Ravenna - Ospedale di Ravenna - IRST, Ravenna
  - Reggio Emilia - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - AUSL della Romagna - Presidio Ospedaliero Rimini - Ospedale "Infermi", Rimini
  - Policlinico Umberto I - Università La Sapienza, Roma
  - Roma - Unicampus-Bio, Roma
  - S. Giovanni Rotondo - Casa Sollievo della sofferenza, San Giovanni Rotondo
  - Siena - Azienda Ospedaliera Universitaria Senese, Siena
  - Terni - Ospedale di Terni, Terni
  - Torino neurooncologia - AOU CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO, Torino
  - Tricase - Ospedale "Card. G. Panico", Tricase
  - Udine, Azienda Ospedaliera Universitaria, Udine
- Switzerland (5):
  - Basel - Universitätsspital, Basel
  - IOSI - Oncology Institute of Southern Switzerland, Bellinzona
  - Bern - Inselspital, Bern
  - St. Gallen - Kantonsspital, Sankt Gallen
  - Universitätsspital Zürich, Zurich